CLINICAL TRIAL: NCT02920554
Title: The Effect in Wedge Resection and IVb/V Resection of the Liver for Gallbladder Cancer Operation: Prospective Randomized Controlled Trial
Brief Title: The Effect in Wedge Resection and IVb/V Resection of the Liver for Gallbladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, YOU DONG DO, Associated Professor, Saint Vincent's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XC14EIMI0009V
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Gallbladder Cancer
Keywords: gallbladder cancer; bisegmentectomy
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- wedge resection (Active Comparator): The extent of hepatic resection is wedge resection of gallbladder fossa
  Interventions: Procedure: wedge resection
- bisegmentectomy (Active Comparator): The extent of hepatic resection is 4b/5 bisegmentectomy
  Interventions: Procedure: bisegmentectomy

INTERVENTIONS:
Procedure: wedge resection — The extent of hepatic resection is wedge resection of liver including gallbladder fossa
  Arms: wedge resection
Procedure: bisegmentectomy — The extent of hepatic resection is 4b/5 bisegmentectomy of liver
  Arms: bisegmentectomy

SUMMARY:
The extent of hepatic resection for gallbladder cancer can be done from a wedge resection to 4b/5 bisegmentectomy. This study aims to compare the recurrence rates and survival rates between wedge resection group and bisegmentectomy group. Patients with T2 or T3 gallbladder cancer on preoperative CT exam or patients who were pathologically diagnosed as T2 or T3 gallbladder cancer after initial simple cholecystectomy were enrolled. All patients are randomly assigned to wedge resection or bisegmentectomy group. Number of patients in each group is 44. Primary endpoint is recurrence-free-survival rates and overall survival rates.

DETAILED DESCRIPTION:
The extent of hepatic resection for gallbladder cancer has a wide range. A partial hepatectomy involving the gallbladder fossa is a critical part of the resection but can range from a wedge resection to an anatomic resection of segments 4b and 5 to an extended right hepatectomy. This study enrolls Patients with T2 or T3 gallbladder cancer on preoperative CT exam or patients who were pathologically diagnosed as T2 or T3 gallbladder cancer after initial simple cholecystectomy. Eighty eight patients are randomized to wedge resection group or bisegmentectomy group. Except the extent of hepatic resection, all the procedures including hepatoduodenal,common hepatic, posterior pancreatic lymph node dissection are same.

Primary endpoint is recurrence-free-survival rates and overall survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2 or T3 gallbladder cancer on preoperative CT exam
* Patients who are pathologically diagnosed as T2 or T3 gallbladder cancer after initial simple cholecystectomy

Exclusion Criteria:

* Peritoneal seeding or distant metastasis
* Impossible to resect the cancer radically
* Pathologically diagnosed to other malignancy such as adenosquamous carcinoma, sarcoma, etc.
* R1 or R2 resection were pathologically diagnosed.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival rates | 1 year
  3year 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Do You, MD, PhD, Study Director — the Catholic Universityof Korea St. Vincent's Hospital
Locations (1):
- the Catholic University of Korea St. Vincent's Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided